CLINICAL TRIAL: NCT01165099
Title: Acupuncture for Pain Relief During Induced Labour in Nulliparae: a Randomised Controlled Study
Brief Title: Acupuncture for Pain Relief During Induced Labour in Nulliparae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Principal Investigator, Ian Mackenzie, Principle investigator, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4874
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Pain
Keywords: acupuncture; induced labour; labour outcome; nulliparae; pain-relief; epidural during labour
MeSH Terms: conditions — Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- manual acupuncture (Experimental): Sterile needles were inserted intramuscularly to a depth of 15-20mm until an unusual (De-Qi) sensation developed and remained inserted for 30-60 minutes and were manually manipulated during this time. The following bilateral acupoints on the hands and feet at Hegu (LI 4), Sanyinjiao (Sp 6) Kunlun (BL 60) and Zhiyin (BL 67)were used.
  Interventions: Procedure: acupuncture
- electro acupuncture (Experimental): Sterile needles were inserted intramuscularly to a depth of 15-20mm until an unusual (De-Qi) sensation developed and remained inserted for 30-60 minutes and were either electronically simulated withm2 Hz pulses of 0.5 msec duration for 30 minutes sufficient to cause non-painful muscle contractions. The following bilateral acupoints on the hands and feet at Hegu (LI 4), Sanyinjiao (Sp 6) Kunlun (BL 60) and Zhiyin (BL 67)were used.
  Interventions: Procedure: acupuncture
- Sham manual or electro acupuncture (Sham Comparator): Sterile needles were inserted adjacent to the specific acupuncture sites identified for the manual and electro groups to a depth of 1-1.5mm only and insufficient to provoke an unusual sensation and left in position for a 30-60 minutes. Those randomised to 'sham-manual' received no stimulation and those randomised to 'sham-electro' were connected to the electrical stimulator but the current not activated.
  Interventions: Procedure: acupuncture
- control group (No Intervention): Following randomisation to be control group, no specific treatment was organised at this time.

INTERVENTIONS:
Procedure: acupuncture — The description of the acupuncture, whether manual, electro or sham, is as described for each of the individual groups.
  Other Names: Disposable needles Seirin DN04 0.20x30mm - 0.30x50mm.; Electronic Acupunctuscope AWQ-104L digital.
  Arms: Sham manual or electro acupuncture; electro acupuncture; manual acupuncture

SUMMARY:
The study was primarily designed to assess the role of acupuncture in reducing the need for epidural analgesia for pain relief during induced labour. The other outcomes of labour were to be observed in addition.

DETAILED DESCRIPTION:
The study was limited to women in their first pregnancy having labour induced for prolonged pregnancy or mild hypertension. The study involved randomised groups managed with manual acupuncture, electro acupuncture, sham acupuncture and a no-treatment control group.

ELIGIBILITY:
Inclusion Criteria:

* nulliparae
* having labour induced for prolonged pregnancy or mild hypertension
* no previous experience of acupuncture
* give written informed consent

Exclusion Criteria:

* all who do not meet the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2005-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
the rate of intrapartum epidural analgesia | within 72 hours of trial entry
  epidural analgesia administered during labour

SECONDARY OUTCOMES:
the outcome of labour | within 72 hours of trial entry
  the outcomes of labour included: parenteral analgesia requirement, labour length, delivery mode, neonatal condition and postpartum haemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: I Z MacKenzie, FRCOG, Principal Investigator — University of Oxford
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom

REFERENCES:
- [Background] Lee H, Ernst E. Acupuncture for labor pain management: A systematic review. Am J Obstet Gynecol. 2004 Nov;191(5):1573-9. doi: 10.1016/j.ajog.2004.05.027. PMID 15547526
- [Result] Mackenzie IZ, Xu J, Cusick C, Midwinter-Morten H, Meacher H, Mollison J, Brock M. Acupuncture for pain relief during induced labour in nulliparae: a randomised controlled study. BJOG. 2011 Mar;118(4):440-7. doi: 10.1111/j.1471-0528.2010.02825.x. Epub 2011 Jan 18. PMID 21244615